CLINICAL TRIAL: NCT03074448
Title: Aquanet Bowel Cleansing Device Versus Oral Sodium Picosulfate for Pre-endoscopy Bowel Preparation: Propensity Score Analysis for Interventional Effectiveness Evaluation
Brief Title: Aquanet Bowel Cleansing Device Versus Oral Sodium Picosulfate for Pre-endoscopy Bowel Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kaiser CH
Record Dates: First submitted 2016-04-25; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Bowel Preparation
Keywords: Colonoscopy; Intestinal Cleaning; Picoprep; Aquanet
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Picosulfate solution (Picoprep) (Active Comparator): On the eve of the examination, all participants on Sodium picosulfate will take four tablets of Dulcolax with tea or water in the morning, liquid diet (juice, tea or water) at lunch, two capsules of 25mg Dramamine Capsgel in the afternoon, Sodium picosulfate dissolved in 150mL of cold water thirty minutes after, followed by drinking at least five 250-ml cups of water or other light liquids until midnight, with absolute fasting up to the time when the colonoscopy will be performed.
  Interventions: Drug: Sodium Picosulfate
- Aquanet bowel cleansing devices (Experimental): For bowel preparation with the bowel cleansing device, intestinal lavage will be performed with the device, making use of water, pressure, and gravity to enhance bowel cleansing. The water used in this procedure was previously triple-filtered by passage on carbon, micro-pellets and ultraviolet light. The preparation will be carried out by a trained nurse.
  Interventions: Device: Aquanet

INTERVENTIONS:
Device: Aquanet — Aquanet bowel cleansing devices
  Arms: Aquanet bowel cleansing devices
Drug: Sodium Picosulfate — Sodium Picosulfate solution (Picoprep)
  Arms: Sodium Picosulfate solution (Picoprep)

SUMMARY:
Poor or inadequate bowel preparation is one of the most common reasons for a repeated or failed colonoscopy. Preparation methods shown to be effective include the use of either bowel-cleansing devices or oral laxatives. Despite the acceptable effectiveness and safety of both bowel-cleansing methods, very few studies have been performed to evaluate which method is more effective. The main aim is to perform an observational study followed by propensity score modeling to evaluate and compare the quality of bowel preparation with the use of Aquanet bowel-cleansing devices versus the use of oral Sodium picosulfate solution. The study will involve 314 patients requiring a colonoscopy, between 14 and 90 years of age and with more than three bowel movements per week for the past one month. Outcomes of interest being the quality of bowel preparation evaluated through the Boston Bowel Preparation (BBP) scale. The investigator hypothesized that the bowel preparation with Aquanet bowel-cleansing device for colonoscopy will provide a better outcome for the patient than with conventional methods.

DETAILED DESCRIPTION:
The study will compare the quality of pre-endoscopic bowel preparation using a bowel-cleansing device with oral Sodium picosulfate solution. The study will be described in accordance with the STROBE (Strengthening the Reporting of Observational studies in Epidemiology) guidelines.

Ethical aspects: The study will undergo full review by the local Institutional Review Board, all potential participants being provided with informed consent. Study protocol will only be initiated after consent is signed.

Settings: Data will be collected from June 2014 to February 2015 at the Portuguese Charitable Hospital, located in Sao Jose do Rio Preto/SP, Brazil. The Kaiser clinic, a private institution, will pay for the Aquanet devices. The Aquanet devices were designed and tested by Prime Pacific Health Innovations Corporation (http://www.primepacifichealth.com/aquanet-family-of-colon-hydrotherapy-devices/), and approved by the various regulatory authorities for market approval and licensing including FDA , Health Canada, and the European Union (<http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPMN/pmn.cfm?ID=K000031>, last accessed October 2016). The Aquanet devices have been on the market since 2001. The procedure lasts for 40-60 min, using filtered, ultraviolet treated water. Water pressure is derived from gravity or from a pump with an upper safe limit of two psi (per square inch) of pressure inside the colon. The device cleanses the large bowel through a series of fill and empty cycles by hydrating the colon, stimulating peristalsis and evacuating bowel contents. The process keeps the body hydrated without losing electrolytes. No adverse events have been reported for the Aquanet devices and there have also been no complaints received to its safety. It may cause mild abdominal discomfort during water infusion in some patients.

Participants: Inclusion criteria will involve all patients requiring a colonoscopy, those between 14 and 90 years of age, and with more than three bowel movements per week for the past one month. Patients will be excluded with following conditions: Pregnancy (confirmed by a pregnancy test), acute abdomen syndrome, prior colorectal surgery, hemorrhoids or endoscopic procedures, known bowel diseases (colon cancer history, toxic megacolon, toxic colitis, idiopathic pseudo obstruction, hypo-motility syndrome), other gastrointestinal disorders (active ulcer, output obstruction, retention, gastroparesis, ileus), previous upper gastrointestinal surgery (gastrectomy, gastric band, gastric bypass), uncontrolled angina and/or myocardial infarction (MI) within the last three months, congestive heart failure (CHF) or uncontrolled hypertension, renal impairment (serum, creatinine and potassium must be within normal limits) or known hypersensitivity to active ingredients. A total of 314 patients will be part of this analysis.

Outcome variables: Major outcome of interest will be the quality of bowel preparation as measured through the Boston Bowel Preparation (BBP) scale. Bowel preparation will be evaluated in three segments: The right segment (cecum and ascending colons), transverse segment (transverse colon including liver and splenic angles), and the left segment (descending and sigmoid colons and rectum). Each segment will be evaluated on a scale from 0-3, and the final score for an individual was the sum of scores for all three segments. Using this score, 0 was the minimum score corresponding to an unprepared colon and 9 was the maximum score corresponding to an excellent preparation without any residual traces.

Predicting variables: Main predictor will be the methods of bowel preparation. The bowel preparation will be done using either Sodium picosulfate or the bowel-cleansing device. On the eve of the examination, all participants on Sodium picosulfate will be given four tablets of Dulcolax with tea or water in the morning, liquid diet (juice, tea or water) at lunch, two capsules of 25mg Dramamine Capsgel in the afternoon, Sodium picosulfate dissolved in 150mL of cold water thirty minutes after, followed by drinking at least five 250-ml cups of water or other light liquids until midnight, with absolute fasting up to the time when the colonoscopy will be performed. For bowel preparation with the bowel cleansing device, intestinal lavage will be performed with the device, making use of water, pressure, and gravity to enhance bowel cleansing. The water used in this procedure will be previously triple-filtered by passage on carbon, micro-pellets and ultraviolet light. The preparation will be carried out by a trained nurse. All endoscopic procedures will be performed by an endoscopist who will be blinded to the method of preparation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 14-90 years
* Must have had >3 spontaneous bowel movements per week for one month prior to the colonoscopy.
* Willing and able to complete the entire process, comply with study instructions, and understand and sign the informed consent.

Exclusion Criteria:

* Pregnancy (women of childbearing age underwent a pregnancy test at screening and again at randomization).
* Acute abdominal surgical conditions (acute obstruction or perforation).
* Prior colorectal surgery (excluding appendectomy), hemorrhoid surgery or endoscopic procedures.
* Bowel disease (colon cancer history, toxic megacolon, toxic colitis, idiopathic pseudoobstruction, hypomotility syndrome).
* Gastrointestinal disorders (active ulcer, output obstruction, retention, gastroparesis, ileus).
* Upper gastrointestinal surgery (gastrectomy, gastric band, gastric bypass).
* Uncontrolled angina and/or myocardial infarction (MI) within the last 3 months; congestive heart failure (CHF) or uncontrolled hypertension.
* Renal impairment (serum, creatinine and potassium must be within normal limits).
* Participation in a research study within 30 days before receiving the study medication (or within 60 days for investigation of drugs with a half-life disposal of more than 15 days).
* Hypersensitivity to active ingredients.
* Chronic kidney disease.
* Latex allergy

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | 16 weeks
  Evaluated through the Boston Bowel Preparation (BBP) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Luiz kaiser Júnior, MD, PhD, Principal Investigator — Kaiser Clinica and Day Hospital
Locations (1):
- Kaiser Clinica and Day Hospital, São José do Rio Preto, São Paulo, Brazil